CLINICAL TRIAL: NCT03291522
Title: Retrieval of Sperm From Men With Azoospermia Using Ultrasound-guided Rete Testis Aspiration
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Infertility and IVF Center, St. Louis, MO (Other)
Responsible Party: Principal Investigator, Kyle Orwig, Professor, University of Pittsburgh
Other Study IDs: PRO17020423
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Azoospermia, Nonobstructive; Infertility, Male
Keywords: Testicular sperm extraction
MeSH Terms: conditions — Azoospermia, Nonobstructive; Infertility, Male

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Men with azoospermia: Ultrasound-guided rete testis flushing and aspiration
  Interventions: Procedure: Ultrasound-guided rete testis flushing and aspiration

INTERVENTIONS:
Procedure: Ultrasound-guided rete testis flushing and aspiration — Ultrasound-guided rete testis flushing and aspiration is performed first. If no sperm is found, the patient can choose to do a standard of care procedure (but not required).

SUMMARY:
The objective of this study is to use ultrasound-guided rete testis flushing and aspiration technique to retrieve sperm, non-surgically, from the testes of azoospermic men. If sperm are retrieved by this method, it will provide a direct benefit to the infertile men. This protocol will also establish the safety and feasibility of the ultrasound-guided rete testis injection approach in consenting men before the approach is translated to teenage boys.

DETAILED DESCRIPTION:
The aim of this study is to demonstrate that ultrasound-guided rete testis aspiration is a safe and effective method to flush and aspirate rare sperm from the testes of men with azoospermia (no sperm in the ejaculate). Current methods to recover sperm from men with azoospermia range from invasive and time consuming micro testicular sperm extraction (microTESE) to fine needle aspiration (FNA), which is less invasive and less time consuming, but also less effective because it is a blind approach. This approach is less invasive; it involves the percutaneous insertion of a hypodermic needle into the rete testis space. This approach is also not blind because the needle is accurately positioned under ultrasound guidance into the rete testis space that is contiguous with all seminiferous tubules (where sperm are made). The investigators will first perform the experimental ultrasound-guided rete testis flushing and aspiration on both testis. If sperm is found, no standard of care procedure (TESE, microTESE etc) will be performed. If sperm is not found, the participant can choose whether or not to proceed with a standard of care procedure. In cases were participants have previously tried a standard of care procedure, they may not want to do that again if the experimental procedure does not work. For the ultrasound-guided rete testis flushing and aspiration, the investigators will flush and aspirate the tubules with 500ul of physiological saline and Optison ultrasound contrast agent in sterile 0.9% saline (routinely used in clinics). Presence of sperm in the aspirate will be determined. The investigators hypothesize that sperm recovery using the ultrasound-guided rete testis injection/aspiration approach will at least as effective as the standard of care approach employed in the Magee male fertility clinic and it will be less invasive.

ELIGIBILITY:
Inclusion Criteria:

* Be a male over the age of 18
* Be diagnosed with azoospermia
* Have 2 testicles
* Sign an approved consent and authorization permitting the release of personal health information. The patient must acknowledge in writing that consent for sperm collection has been obtained, in accordance with institutional policies approved by the U.S. Department of Health and Human Services.

Exclusion Criteria:

* Diagnosed with psychological, psychiatric, or order conditions which prevent giving fully informed consent
* Diagnosed with underlying medical condition that significantly increases their risk of complications from this procedure

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males over the age of 18 who are diagnosed with azoospermia.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-05-10 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Presence of sperm | 5 years
  Percentage of time that sperm is found with ultrasound-guided rete testis aspiration

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Orwig, PhD, Principal Investigator — University of Pittsburgh/University of Pittsburgh Medical Center
Locations (1):
- Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided